CLINICAL TRIAL: NCT00459030
Title: Two Delivery Channels to Improve CRC Screening
Brief Title: Traditional Print Communication Methods, Simple Electronic Communication Methods, or Usual Care in Increasing How Often Older Women Undergo Colorectal Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FCCC-05016; CDR0000538413 (Registry Identifier: PDQ (Physician Data Query)); IRB05-016 (Other: Fox Chase Cancer Center); R01CA102695 (NIH)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Print Communication (Experimental): Cancer screening educational information mailed to patient's home one time after signing consent.
  Interventions: Other: educational intervention mailed
- Electronic communication (Experimental): Cancer screening educational information delivered via a password protected internet site.
  Interventions: Other: educational intervention via internet
- No Health Communication (Active Comparator): No additional cancer screening education information sent to patient.
  Interventions: Other: No additional educational intervention

INTERVENTIONS:
Other: educational intervention via internet — additional cancer screening information via password protected internet site
  Arms: Electronic communication
Other: educational intervention mailed
  Arms: Print Communication
Other: No additional educational intervention
  Arms: No Health Communication

SUMMARY:
RATIONALE: Finding out which communication method affects a participant's decision to undergo colorectal cancer screening may help increase the number of participants who undergo screening. It is not yet known which communication method is more effective in increasing how often participants undergo colorectal cancer screening.

PURPOSE: This randomized clinical trial is studying traditional print communication methods to see how well they work compared with simple electronic communication methods or usual care in increasing how often older women undergo colorectal cancer screening.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare traditional print versus simple electronic communication versus usual care, in terms of increasing colorectal cancer (CRC) screening rates, in average-risk women attending a routine OB/Gyn visit.
* Explore the moderating role of attentional style and background variables on the impact of the interventions in these participants.
* Determine the mediating effect of potential cognitive-affective factors related to CRC screening in these participants.
* Investigate the comparative cost-effectiveness of these interventions to improve CRC screening adherence.

OUTLINE: This is a randomized study. Participants are randomized to 1 of 3 screening arms.

* Arm I: Participants are contacted by simple electronic communication methods by an email message linked to a personalized website.
* Arm II: Participants are contacted by traditional print communication methods.
* Arm III: Participants are observed (usual care). Participants in arms I and II are randomized a second time to receive messages about colorectal cancer screening that are matched or mismatched to their attentional style.

PROJECTED ACCRUAL: A total of 5,000 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At average risk for colorectal cancer (CRC) as defined by the following criteria:

  * Asymptomatic without a personal history of colorectal polyps or cancer
  * No inflammatory bowel disease
  * No family history of familial adenomatous polyposis or hereditary nonpolyposis CRC
  * No CRC in more than one first-degree relative
* Nonadherent with standard CRC screening recommendations at the time of index OB/Gyn appointment

PATIENT CHARACTERISTICS:

* Email accessible at home and/or work
* Able to communicate with ease in English

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 904 (Actual)
Dates: Start 2005-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Comparison of traditional print versus simple electronic communication versus usual care in terms of increasing colorectal cancer (CRC) screening rates | End of study

SECONDARY OUTCOMES:
Moderating role of attentional style and background variables on the impact of the interventions | End of Study
Mediating effect of potential cognitive-affective factors related to CRC screening | End of study

CONTACTS AND LOCATIONS:
Overall Officials: David Weinberg, MD, MSC, Study Chair — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Weinberg DS, Keenan E, Ruth K, Devarajan K, Rodoletz M, Bieber EJ. A randomized comparison of print and web communication on colorectal cancer screening. JAMA Intern Med. 2013 Jan 28;173(2):122-9. doi: 10.1001/2013.jamainternmed.1017. PMID 23128366